CLINICAL TRIAL: NCT06109519
Title: A Comparative Clinical Study for Two Types of Locator Attachments for Mandibular Implant-supported Overdenture; A 3-year Radiographic and Clinical Follow-up Study
Brief Title: Comparative Clinical Study for Two Types of Locator Attachments for Mandibular Implant Supported Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0208023RP
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Prosthesis User

STUDY DESIGN:
Intervention Model Description: All patients in this study will be divided into two equal groups Group I (control): patients who would be delivered mandibular implant overdenture using conventional locator attachments.
  Group II (study): patients who would be delivered mandibular implant overdenture using Locator RTX attachments
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): patients who would be delivered a mandibular implant overdenture using conventional locator attachments.
  Interventions: Procedure: implant supported overdenture
- Group II (study) (Active Comparator): patients who would be delivered mandibular implant overdenture using Locator RTX attachments
  Interventions: Procedure: implant supported overdenture

INTERVENTIONS:
Procedure: implant supported overdenture — patients would be delivered mandibular implant overdenture using conventional locator and Locator RTX attachments

SUMMARY:
This study aims to evaluate the clinical and radiographic outcomes for mandibular implant-supported overdenture using two different types of locator attachment after 3 years of using the two types of locator attachments

ELIGIBILITY:
Inclusion Criteria:

* 1. All selected patients have two implants placed in the mandibular interforaminal region.

  2. All selected patients have a healthy mucosa and with no clinical complications.

  3. All patients are cooperative and approve the proposed treatment protocol

Exclusion Criteria:

* 1. Patients who reject to participate in the study. 2.Patients who need implant placement as a result of previous implant failure

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-16 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2023-09-16 (Actual)

PRIMARY OUTCOMES:
crestal cone loss | three years
  Intraoral radiographs were performed using the long cone paralleling technique to evaluate crestal bone loss
prosthetic complications | three years
  prosthetic complications were scored clinically

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University ,Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No